CLINICAL TRIAL: NCT01691066
Title: Pivotal Response Treatment for Infants At-Risk for Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1110009256; R03MH092617 (NIH)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

ARMS (2):
- Infant Toddler Years PRT (Experimental): Infant Toddler PRT in an evidence-based, manualized treatment for children with autism spectrum disorder that involves specific motivational behavioral procedures adapted to be developmentally appropriate for 12-15 month old infants who present with developmental delays.
  Interventions: Behavioral: Infant Toddler Years PRT
- Community Treatment (No Intervention): Community Treatment includes the treatments offered by early intervention services (e.g., speech-language therapy, special education instruction).

INTERVENTIONS:
Behavioral: Infant Toddler Years PRT
  Other Names: Pivotal Response Treatment
  Arms: Infant Toddler Years PRT

SUMMARY:
The purpose of this study aims to investigate the utility of Pivotal Response Treatment (PRT), a behaviorally derived intervention, to improve the quality and frequency of communication and social engagement of toddlers with siblings who have an autism spectrum disorder (SIBS - ASD) and who demonstrate developmental delays and impairments in social interaction between 12 and 15 months of age.

ELIGIBILITY:
Inclusion Criteria:

* toddlers, age 12 - 15 months, who have an older sibling with ASD
* delays of at least 1.5 standard deviations in communication (receptive/expressive language) based on developmental testing
* scores that exceed the ASD cutoff on standardized measures of social-communicative behavior

Exclusion Criteria:

* physical or neurological disorder (e.g., seizures, cerebral palsy)

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of a novel behavioral treatment | 24 months
  Assessment of Outcome:
  Attendance. Attendance to parent education sessions will be recorded by the therapist.
  Parent utilization. To assess the acceptability of the PRT approach, parents will be asked to keep a weekly log of procedure use, including overall estimated duration and choice of activities.
Acceptability of a novel behavioral treatment | 24 months
  Assessment of Outcome:
  Parent satisfaction. At post-treatment, parents will be asked to complete a Likert-scale and short response questionnaire rating their satisfaction with various aspects of the program

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Chawarska, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States